CLINICAL TRIAL: NCT04217408
Title: Deep Brain Stimulation (DBS) of the Ventral Capsule/Ventral Striatum (VC/VS) for the Treatment of Refractory Obsessive-compulsive Disorder (OCD)
Brief Title: Deep Brain Stimulation (DBS) for the Treatment of Refractory Obsessive-compulsive Disorder (OCD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Dr Nir Lipsman, MD, PhD, Neurosurgeon, Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111-2018
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: 1 year of open-label treatment, followed by 5 week double blinded crossover phase consisting of 2 weeks of ON stimulation and 2 weeks of OFF stimulation separated by a 1 week washout period with OFF stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent member of the study team will perform the randomization and programming, allow for care givers, participants, investigator, and outcomes assessors to be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ON stimulation followed by OFF stimulation (Experimental): All patients complete the same 52 week open-label phase with active stimulation. After this, they enter a blinded randomized crossover phase of 2 weeks of ON (active) stimulation, followed by 2 weeks of OFF (sham) stimulation
  Interventions: Device: Deep brain stimulation
- OFF stimulation followed by ON stimulation (Experimental): All patients complete the same 52 week open-label phase with active stimulation. After this, they enter a blinded randomized crossover phase of 2 weeks of OFF (sham) stimulation, followed by 2 weeks of ON (active) stimulation
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Active continuous deep brain stimulation of the ventral capsule/ventral striatum

SUMMARY:
Deep brain stimulation for treatment resistant deep brain stimulation

DETAILED DESCRIPTION:
Subjects will receive bilateral deep brain stimulation to the ventral capsule/ventral striatum. They will receive standard follow-up and device programming over the span of 52 weeks. After that, they will enter a 5 week double blinded crossover phase consisting of 2 weeks of ON or OFF stimulation, separated by 1 week of 'washout', during which stimulation will be OFF.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male patients between age 18-70
2. DSM-V diagnosis of Obsessive Compulsive Disorder (OCD), at least 5-year illness history with a minimum score of 24 on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS).
3. SF-36<40
4. Medication-refractoriness as determined by an adequate dose and duration of psychiatric treatments (including psychotherapy and/or pharmacology) as determined by two psychiatrists associated with the study. Including specifically:

   1. Failed adequate trial of two or more medications accepted as first line in the treatment of OCD
   2. Attempted augmentation, if tolerated, by at least 1 medications known to be first line treatments for OCD
5. An adequate trial of cognitive behavioural therapy
6. Ability to provide informed consent and comply with all testing, follow-ups and study appointments and protocols

Exclusion Criteria:

1. Any past or current evidence of psychosis or mania (patients with co-morbid depression will not be excluded from the study)
2. Active neurologic disease, such as epilepsy
3. Alcohol or substance dependence or abuse in the last 6 months, excluding caffeine and nicotine
4. Current suicidal ideation
5. Any contraindication to MRI scanning
6. No contraindication for DBS surgery
7. Presence of significant cognitive impairment
8. Likely to relocate or move out of the country during the study's duration
9. Presence of clinical and/or neurological conditions that may significantly increase the risk of the surgical procedure.
10. Currently pregnant (as determined by history and serum HCG) or lactating; for females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-12-19 (Estimated); Study Completion 2024-12-19 (Estimated)

PRIMARY OUTCOMES:
Quality of Life as measured by the Short-Form 36 | 12 months compared to baseline
  Measured by the short form 36 (SF-36). The scores range from 0-100 with lower numbers indicating a worse quality of life.

SECONDARY OUTCOMES:
Obsessive compulsive symptoms as measured by the Yale-Brown Obsessive Compulsive Scale | 12 months
  Change in Yale-Brown Obsessive Compulsive Scale score at 12 months compared to baseline. The scores range from 0-40, with high scores indicating more severe obsessions and compulsions.
Obsessive compulsive symptoms as measured by the Yale-Brown Obsessive Compulsive Scale during randomization | Recorded at the end of the 2 week ON and OFF stimulation periods, which occur immediately after the 52 week open-label period
  Yale-Brown Obsessive Compulsive Scale score during active ON stimulation compared to during OFF stimulation. The scores range from 0-40, with high scores indicating more severe obsessions and compulsions.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided